CLINICAL TRIAL: NCT02561117
Title: Metronidazole Every 24 Hours as Part of Triple Antibiotic Therapy for Ruptured Appendicitis in Children Managed Operatively (METRO): a Noninferiority Randomized Controlled Trial
Brief Title: Once Daily Metronidazole for Perforated Appendicitis
Acronym: METRO
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Ahmed Nasr (Other)
Responsible Party: Sponsor-Investigator, Ahmed Nasr, Principal Investigator, Children's Hospital of Eastern Ontario
Organization: Children's Hospital of Eastern Ontario (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4660
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- q8h (Active Comparator): Metronidazole given every 8 hours
  Interventions: Drug: Metronidazole
- q24h (Experimental): Metronidazole given once daily
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — Administration once daily
  Other Names: Flagyl

SUMMARY:
The objective of this study is to determine whether administering once-daily doses of metronidazole, an intravenous (IV) antibiotic used to prevent infection in perforated appendicitis, is as effective in children as delivering it in the standard method of once every eight hours. Reducing the frequency of administration has the potential of decreasing personnel time and healthcare cost and increasing the lifespan of the IV line.

To determine the effectiveness once-daily administration, a randomized controlled trial (RCT) will be conducted to compare outcomes between the two treatment schedules. We will recruit 100 patients (50 per treatment) aged 5-18 being surgically treated for perforated appendicitis at the Children's Hospital of Eastern Ontario, who will be randomly assigned to one of the two treatment schedules. To compare the efficacy of the treatments, outcomes such as duration of hospital stay and theoretical cost will be measured and analyzed using statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* All children 5-18 years of age, presenting to CHEO with perforated appendicitis (confirmed either in the operating room or diagnosed preoperatively according to radiological criteria), and managed surgically will be assessed for eligibility to participate. These patients may participate if baseline lab values of serum AST (SGOT), AL T (SGPT), LDH, triglycerides and hexokinase glucose are normal, complete physical exam is normal, hGC test is negative for pregnancy (if the patient is a female of reproductive age) and none of the exclusion criteria are present.

Exclusion Criteria:

* Any known co-existing gastrointestinal disease
* Uncertainty about the diagnosis
* Perforated appendicitis with diffuse abdominal fluid on imaging associated with a clinical picture of severe sepsis
* A known allergy to any of the antibiotics to be used in this trial
* An active neurological disorder
* Receiving medical treatment for a neurological disorder
* A history of blood dyscrasia, hypothyroidism or hypoadrenalism
* Hepatic disease
* Renal impairment
* Patients receiving any other oral or intravenous concomitant antimicrobial at enrollment
* Pregnancy
* Under five years of age
* Patients who have received metronidazole orally or intravenously in the last 14 days, prior to the current admission for appendicitis
* Patients already taking any of the following medications at admission (as these may interact with Metronidazole as stated in the product monograph): disulfiram, oral anticoagulant therapy (warfarin type), phenytoin or phenobarbital, vecuronium, lithium, busulfan
* The physician elects to treat the patient conservatively (non-surgically)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Length of stay | until discharge (usually less than one week after admission)
  • Duration of hospital stay (in days) during initial admission for perforated appendicitis (Patient will be discharged when eating normal diet, afebrile for 24 hours and no abdominal pain)

SECONDARY OUTCOMES:
Failure of antibiotics | during hospital stay (usually less than one week)
  o No clinical improvement after five days, as decided by the patient's surgeon. This will result in the patient being switched to a regimen of different antibiotics.
Quantity of narcotics | From date of randomization to date of death from any cause or three months after initial discharge from hospital, whichever comes first.
  mg/kg per day of narcotics
Duration of narcotics | From date of randomization to date of death from any cause or three months after initial discharge from hospital, whichever comes first.
  total number of days of narcotics
Duration of antibiotics IV | From date of randomization to date of death from any cause or three months after initial discharge from hospital, whichever comes first.
  duration of IV antibiotic therapy (days)
Duration of antibiotics oral | From date of randomization to date of death from any cause or three months after initial discharge from hospital, whichever comes first.
  duration of oral antibiotic therapy following discharge (days)
Theoretical cost in CAD | From date of randomization to date of death from any cause or three months after initial discharge from hospital, whichever comes first.
  In our study, due to blinding, much of the potential cost-savings of once-daily administration of metronidazole - including nursing time, pharmacy time, and IV materials - will not be evident. However, we will calculate the potential cost-savings of once-daily administration. This will be based on number of hours of nursing time saved (the research coordinator (RC) will, on 10 occasions, observe a nurse administering a dose of metronidazole to a patient not enrolled in this study, and will average these to estimate the time required to administer one dose), number of hours of pharmacy time saved (the RC will, on 10 occasions, observe a pharmacist preparing a dose of metronidazole for a patient not enrolled in this study, and will average these to estimate the time required to prepare one dose), and cost saved on materials (the minibag used to deliver the antibiotic, the IV needle and line if it needed to be replaced, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Nasr, Principal Investigator — CHEO